CLINICAL TRIAL: NCT05320627
Title: Population Pharmacokinetics of Edoxaban in Chinese Patients With Non-Valvular Atrial Fibrillation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EPP-AF-102
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Non-Valvular Atrial Fibrillation
Keywords: Edoxaban; Population Pharmacokinetics; Non-Valvular Atrial Fibrillation
MeSH Terms: interventions — edoxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Edoxaban treatment (Experimental)
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Eligible patients will receive Edoxaban tablet once a day for 12 weeks

SUMMARY:
Based on the population pharmacokinetic data of Chinese patients with atrial fibrillation, the study will evaluate the suitability of the ENGAGE Population Pharmacokinetics model of edoxaban in patients with atrial fibrillation in China, and build a predictive dose model of edoxaban that meets the characteristics of Chinese people. It can provide perfect individualized dosing plan improves clinical efficacy and reduces adverse drug reactions.

DETAILED DESCRIPTION:
This is an open label study. Male or female patients with non-valvular atrial fibrillation (NVAF) with age ≥20 years, and meeting the indications of edoxaban are potentially eligible for the study. Patients receive Edoxaban 15mg、30mg or 60mg according to the criteria as following:

1. Patients with severe renal insufficiency (15ml/min ≤ CrCl <30ml/min), 15mg quaque die (QD)
2. Patients with normal or mild renal insufficiency (CrCl ≥50ml/min), 60mg QD
3. Patients with moderate renal insufficiency (30ml/min ≤ CrCl <50ml/min), weight ≤60kg or combined use of P-gp inhibitors (such as dronedarone，ketoconazole, erythromycin, etc), 30mg QD.

Patients will receive clinical evaluation at screening period, 4 weeks、8 weeks and 12 weeks after administration with Edoxaban. The following clinical evaluation items were included: body weight, vital signs (blood pressure and heart rate), CHADS2-VAS score, concomitant medication, ECG and echocardiogram, laboratory examination, safety evaluation (thromboembolic events, bleeding events, death) during treatment.

Additional blood samples are collected for pharmacokinetic evaluation at screening period, pre-dose, 2±1h and 6±1h after administration at 4-, 8-, and 12-week visit, and for pharmacodynamic evaluation (FXa) at screening period, pre-dose after administration at 4-, 8-, 12-week visit.

The population pharmacokinetics of Edoxaban in Chinese patients with non-valvular atrial fibrillation will be determined after 12weeks clinical observation.

The ENGAGE PopPK model suitable in Chinese Patients with Non-Valvular Atrial Fibrillation will be established.

Safety outcomes (thromboembolic events, bleeding events, death) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female NVAF patients, who need anticoagulant therapy at least 3 months
2. Age ≥20 years,
3. Creatinine clearance rate ≥ 15 ml/min
4. Sign a written informed consent form (ICF) for participating in the study
5. No simultaneous participation in any interventional study

Exclusion Criteria:

1. Patients with the Valve replacement
2. Patients with valvular atrial fibrillation
3. Mild and severe anemia patients
4. CrCl<15ml/min
5. Patients on dialysis, risk of bleeding, taking antiplatelet drugs, or taking other anticoagulants
6. Contraindicated to Edoxaban.
7. Life expectancy < 6 months.
8. Hypertension defined as systolic and/or diastolic blood pressure > 95th age percentile or poorly controlled hypertension
9. Hepatic disease which is associated either: with coagulopathy leading to a clinically relevant bleeding risk, or alanine transaminase (ALT) > 5x upper level of normal (ULN), or total bilirubin > 2x ULN with direct bilirubin > 20% of the total.
10. Active bleeding or high risk for bleeding contraindicating anticoagulant therapy. For example：

    * a history of intracranial, intraocular, intraspinal, retroperitoneal, or traumatic intra-articular bleeding
    * gastrointestinal bleeding during the prior year
    * peptic ulcer within the previous 90 days
    * surgery or injury requiring hospitalization within the previous 30 days
    * hemoglobin <9 g/dl or a platelet count <50×109/L
    * active bleeding at registration
    * any procedure associated with bleeding planned to occur during the treatment period
11. Urine pregnancy test positive if female
12. Inability to cooperate with the study procedures
13. Participation in a study with an investigational drug or medical device within 30 days prior to screening
14. Additional exclusion criteria included, but were not limited to:

    * cerebral infarction or transient ischemic attack within the past 30 days
    * comorbid rheumatic valvular disease
    * comorbid infective endocarditis or atrial myxoma
    * evidence of thrombus in the left ventricle or atrium, or hereditary tendency for thrombus formation scheduled electrical or pharmacological defibrillation during the treatment period
    * acute myocardial infarction, or unstable angina
    * a diagnosis of active malignant tumor or cancer treatment within the past 5 years
    * previous treatment with Edoxaban

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
population pharmacokinetic evaluation | at the 4th, 8th and 12th week
  Patients enrolled will be back to center for visit at scheduled timepoint. Blood sample for PopPK study was collected. Edoxaban concentrations in patient plasma will be determined, which will be analysed and compared with ENGAGE PopPK model.
pharmacokinetic evaluation | at the 4th, 8th and 12th week
  Patients enrolled will be back to center for visit at scheduled timepoint. Blood for pharmacodynamic sample will be collected for Anti-FXa activity determination.

SECONDARY OUTCOMES:
safety evaluation | at the 4th, 8th and 12th week
  Patients enrolled will be back to center for visit at scheduled timepoint. Adverse even will be recorded. The investigator will determine whether the patient is suitable to go on with the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hua, 1, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital; Lei Tian, 2, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No